CLINICAL TRIAL: NCT03797196
Title: Open Label Multicenter Randomized Trial Comparing Standard Immunosuppression With Tacrolimus and Mycophenolate Mofetil With a Low Exposure Tacrolimus Regimen in Combination With Everolimus in de Novo Renal Transplantation in Elderly Patient
Brief Title: RCT Comparing Immunosuppressive Regimens in Elderly Renal Transplant Recipients
Acronym: OPTIMIZE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Radboud University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amsterdam UMC, location VUmc (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); Erasmus Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, principal investigator, head of renal transplant program UMCG, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMIZE
Record Dates: First submitted 2018-12-11; First posted 2019-01-09 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Renal Transplant Recipients; Elderly Patients; Immunosuppression
MeSH Terms: interventions — Tacrolimus; Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator): standard tacrolimus with mycophenolate mofetil
  Interventions: Drug: standard dose tacrolimus with mycophenolate mofetil
- group 2 (Experimental): low dose tacrolimus with everolimus
  Interventions: Drug: low dose tacrolimus in combination with everolimus

INTERVENTIONS:
Drug: low dose tacrolimus in combination with everolimus — a low exposure Tacrolimus once-daily (Envarsus®) regimen in combination with Everolimus will be evaluated in elderly transplant recipients
  Arms: group 2
Drug: standard dose tacrolimus with mycophenolate mofetil — A standard Tacrolimus once-daily (Envarsus) regimen in combination with Everolimus will be evaluated in elderly transplant recipients
  Arms: group 1

SUMMARY:
Open label, randomized, multicenter, intervention trial comparing standard immunosuppression with tacrolimus and mycophenolate mofetil with a low exposure tacrolimus regimen in combination with everolimus.

The primary objective is to test the hypothesis that an age-adapted immunosuppressive regimen targeted at reduced immunosuppression with low calcineurin inhibitor (tacrolimus) exposure in combination with everolimus will result in improved outcome in elderly recipients of A: Kidneys from older deceased donors (>64 years) and B: Kidneys from living donors (all ages) and younger deceased donors (<65 years).

DETAILED DESCRIPTION:
In this study two immunosuppressive regimes will be tested; In both groups basiliximab induction will be applied. Additionally, the standard therapy consisting of prednisolone, mycophenolic acid and tacrolimus once-daily (Envarsus®), or the comparator in which mycophenolic acid will be replaced by everolimus combined with strongly reduced levels of tacrolimus once-daily (Envarsus®). When not tolerated,tacrolimus may be replaced by ciclosporin. The hypothesis is that reduced calcineurin inhibitor (CNI) exposure in combination with everolimus will lead to improved allograft function, a reduced incidence of complications and improved quality of life.

This study will consist of two strata: Stratum A: Elderly recipients (≥65 years) of kidneys from elderly deceased donors (≥65 years) within the Eurotransplant Senior Program. Stratum B: Elderly recipients (≥65 years) of kidneys from living donors (all ages) or deceased donors (<65 years). The primary endpoint will be "successful transplantation" which is defined as survival with a functioning allograft with a minimum estimated GFR of 30 ml/min per 1.73 m2 in stratum A and 45 ml/min per 1.73 m2 in stratum B, after 2 years.

The study will be performed by the Dutch transplant centers and the Dutch Kidney Patient Organization (NVN) will participate.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed
2. Male or female subject ≥65 years old
3. Subject randomized within 24 hours of completion of transplant surgery
4. Stratum A: Recipient of a primary (or secondary, if first graft is not lost due to immunological reasons) renal transplant from a deceased donor aged 65 years or older
5. Stratum B: Recipient of a primary (or secondary, if first graft is not lost due to immunological reasons) renal transplant from a deceased donor aged below 65 years or a living donor of any age

Exclusion Criteria: Exclusion criteria for both stratum A and B

1. Subject is a multi-organ transplant recipient
2. Recipient of bloodgroup ABO incompatible allograft or CDC cross-match positive transplant
3. Subject at high immunological risk for rejection as determined by local practice for assessment of anti-donor reactivity
4. Recipient of a kidney with a cold ischaemia time (CIT) >24 hr
5. Recipients of a kidney from an HLA-identical related living donor
6. Known intolerability for one or more of the study drugs
7. Subject who is HIV positive
8. HBsAg and/or a HCV positive subject with evidence of elevated liver function tests (ALT/AST levels ≥2.5 times ULN). Viral serology results obtained within 6 months prior to randomization are acceptable
9. Recipient of a kidney from a donor who tests positive for human immunodeficiency virus, (HIV), hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV)
10. Subject with severe systemic infections, current or within the two weeks prior to randomization
11. Subject with severe restrictive or obstructive pulmonary disorders
12. Subject with severe hypercholesterolemia or hypertriglyceridemia that cannot be controlled
13. Subject with white blood cell (WBC) count ≤ 2,000/mm3 or with platelet count ≤ 50,000/mm3

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
successful transplantation | 24 months
  The overall primary study endpoint "successful transplantation" as defined for the individual strata and analyzed for the whole study population.
  Stratum A: Primary endpoint: successful transplantation at two years after transplantation defined as: absence of graft or patient loss in the presence of an eGFR above 30 ml/min/1.73m2.
  Stratum B: Primary endpoint: successful transplantation at two years after transplantation defined as absence of graft or patient loss in the presence of an eGFR above 45 ml/min/1.73m2

SECONDARY OUTCOMES:
death | 24 months
  patient survival
graft loss | 24 months
  graft survival
acute rejection | 24 months
  treated biopsy-proven rejection (tBPAR)
eGFR | 12 and 24 months
  estimated Glomerular Filtration Rate below 30 and 45 ml/min/1.73m2
type of rejection treatment | 24 months
  type of rejection treatment will be scored by questionnaire to the treating nephrologist
The evolution of renal function (eGFR) and creatinine clearance over time by slope analysis | 24 months
  The evolution of renal function (eGFR) and creatinine clearance over time by slope analysis
The incidence of adverse events, serious adverse events and adverse reactions | 24 months
  The incidence of adverse events, serious adverse events and adverse reactions
The incidence of clinically relevant infections, post transplantation diabetes mellitus, malignancies and cardiovascular events | 24 months
  The incidence of clinically relevant infections, post transplantation diabetes, malignancies and cardiovascular events
Presence of frailty after transplantation and change in frailty from baseline frailty from baseline | 12 and 24 months
  frailty is measured by clinical frailty score, hand grip strength and fried frailty index
Physical functioning and changes over time | 24 months
  Short Physical Performance Battery
Cognitive functioning and changes over time | 24 months
  Montreal Cognitive Assessment
Presence of T-cell immunosenescence at 12 and 24 months and changes from baseline | 24 months
  T cell differentiation, exhaustion and telomere length will be assessed by flowcytometry
HRQoL at 0, 12 and 24 months and changes from baseline | 24 months
  Questionnaire: EQ-5D and SF-12
Development of donor-specific anti-HLA antibodies (DSA) | 24 months
  DSA as measured by Luminex
Difference in illness perception at 0, 12 and 24 months and changes from baseline | 24 months
  Questionnaire: Brief Illness Perception Questionnaire
Difference in adherence of immunosuppressive medication at 12 and 24 months | 24 months
  Questionnaire: Basel Assessment of Adherence to Immunosuppressive Medication Scale
Difference in symptoms at 0, 12 and 24 months and changes from baseline | 24 months
  Questionnaire: Dialysis Symptom Index with additional items from the Modified Transplant Symptom Occurrence and Symptom Distress Scale-59
Difference in iBOX predicted outcome at 3, 5 and 7 years | 24 months
  Based on the available data
Development of a pharmacokinetic model for tacrolimus once-daily (Envarsus®), using data on AUC's | 24 months
  In addition to trough levels, additional AUC's will be withdrawn at the Leiden University Medical Center as routine patient care on week 2 and 6.
o evaluate the response to the COIVD-19 vaccine and identify possible differences between both treatment groups at the University Medical Center Groningen. | 24 months
  Humoral and T-cell response

OTHER OUTCOMES:
Evaluation of Cost-effectiveness of the new immunosuppressive regimen, and comparison to the current standard of care | 24 months
  Cost-effectiveness of the immunosuppressive regimen will be evaluated using state-of-the-art health-economic techniques; costs and effectiveness of immunosuppressive therapy will be derived from the study

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hesselink, MD, PhD, Principal Investigator — EMC; Frederike Bemelman, Md, PhD, Principal Investigator — AIDS Malignancy Consortium; Stefan Berger, Md, PhD, Study Chair — University Medical Center Groningen; Jan-Stephan Sanders, MD, PhD, Study Director — University Medical Center Groningen; Azam Nurmohamed, Md, PhD, Principal Investigator — VUMC; Aiko De Vries, MD, PhD, Principal Investigator — LUMC; Luuk Hilbrands, Md, PhD, Principal Investigator — Radboud MC; Arjan Van Zuilen, MD, PhD, Principal Investigator — UMCU; Dirk Kuypers, MD, PhD, Principal Investigator — Leuven MC
Locations (7):
- Leuven University Hospital, Leuven, Belgium
- Netherlands (6):
  - Amsterdam UMC, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - Radboud University Hospital, Nijmegen
  - Erasmus MC, Rotterdam
  - UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanders JF, de Boer SE, Jonker J, Bemelman FJ, Betjes MGH, de Vries APJ, Hilbrands L, Hilhorst M, Kuypers DRJ, Vart P, van Zuilen AD, Hesselink DA, Berger SP. Immunosuppression in Older Kidney Transplant Recipients: A Randomized Controlled Trial. J Am Soc Nephrol. 2025 Nov 7. doi: 10.1681/ASN.0000000924. Online ahead of print. No abstract available. PMID 41201871
- [Derived] Oliveras L, Lopez-Vargas P, Melilli E, Codina S, Royuela A, Coloma Lopez A, Fava A, Manonelles A, Couceiro C, Lloberas N, Cruzado JM, Montero N. Delayed initiation or reduced initial dose of calcineurin-inhibitors for kidney transplant recipients at high risk of delayed graft function. Cochrane Database Syst Rev. 2025 Apr 8;4(4):CD014855. doi: 10.1002/14651858.CD014855.pub2. PMID 40197799
- [Derived] de Boer SE, Sanders JSF, Bemelman FJ, Betjes MGH, Burgerhof JGM, Hilbrands L, Kuypers D, van Munster BC, Nurmohamed SA, de Vries APJ, van Zuilen AD, Hesselink DA, Berger SP. Rationale and design of the OPTIMIZE trial: OPen label multicenter randomized trial comparing standard IMmunosuppression with tacrolimus and mycophenolate mofetil with a low exposure tacrolimus regimen In combination with everolimus in de novo renal transplantation in Elderly patients. BMC Nephrol. 2021 Jun 2;22(1):208. doi: 10.1186/s12882-021-02409-8. PMID 34078323